CLINICAL TRIAL: NCT05751252
Title: Short-term GnRH- Antagonist Treatment to Lower LH Pulsatility in Women With PCOS Aiming to Improve Hormonal Functions
Brief Title: Sub-therapeutic GnRH- Antagonist Treatment to Rectify LH Pulsatility in Lean Women With PCOS.
Acronym: SOPKGANI
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022_0016; 2023-000176-35 (EudraCT Number)
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; GnRH antagonist; LH; androgen; testosterone
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.0625 mg (Experimental): Test the efficacy of Ganirelix administered subcutaneously at single-dose regimen of 0.0625 mg in 10 women with PCOS, in rectifying LH pulse frequency and LH amplitude
  Interventions: Drug: Ganirelix
- 0.025 mg (Experimental): Test the efficacy of Ganirelix administered subcutaneously at single-dose regimen of 0.025 mg in 10 women with PCOS, in rectifying LH pulse frequency and LH amplitude.
  Interventions: Drug: Ganirelix

INTERVENTIONS:
Drug: Ganirelix — An intra-venous cannula will be inserted and blood will be sampled at 10-min intervals for a 4-h baseline period commencing at 0800 h. Ganirelix will be then administered subcutaneously at single-dose regimen at 0.0625 mg (n = 10 women with PCOS). After Ganirelix administration sampling will continue at 10-min intervals for 4 h.
  Arms: 0.025 mg
Drug: Ganirelix — An intra-venous cannula will be inserted and blood will be sampled at 10-min intervals for a 4-h baseline period commencing at 0800 h. Ganirelix will be then administered subcutaneously at single-dose regimen at 0.025 mg (n = 10 women with PCOS). After Ganirelix administration sampling will continue at 10-min intervals for 4 h.
  Arms: 0.0625 mg

SUMMARY:
The clinical study using a sub-therapeutic dose of a GnRH antagonist to reduce overactive LH pulsatility in women with PCOS. With the intervention and lowered LH action we anticipate to decrease androgen levels in women with PCOS. The aim to show for the first time that low-dose GnRH-antagonists can lower LH pulsatility by 20-30% and decrease androgen levels without blunting the hypothalamic-pituitary-gonadal axis and thereby the reproductive functions.

ELIGIBILITY:
Inclusion Criteria:

* Minimum weight of 51 kg
* BMI between 20 and 25
* women with PCOS with AMH> 28 pmol / L, LH> 8 IU / mL and testosteronemia > 0.39 ng/mL
* no hormonal treatment or contraception for 2 months
* women covered by the Social Security system

Exclusion Criteria:

* hormonal treatment or hormonal contraception
* Metformin treatment
* pregnant woman
* inability to understand the newsletter

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients followed in endocrine gynecology consultation in the Jeanne de Flandre department
Enrollment: 20 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-02-09 (Actual); Study Completion 2025-02-09 (Actual)

PRIMARY OUTCOMES:
Serum LH level | every 10 minutes for 8 hours
  The degree of gonadotropin suppression will be determined by calculating the percent inhibition from the pre-antagonist period [(mean PRE - nadir)/mean PRE] x 100, where nadir hormone levels will be calculated using a moving average.

SECONDARY OUTCOMES:
Variation in LH secretion amplitude before and after Ganirelix* injection (area under the curve) | at the beginning and at the end of the 8 hours
Variation in androgen production | at 4 hours after injection
  defined by the difference between the measurement at H8 and the measurement at H0 (4 hours before injection) of total testosterone and androstenedione.
change in FSH levels | at 4 hours post-injection
  defined as the difference between the measurement at H8 and the measurement at H0 (4 hours prior to injection) of FSH
change in estradiol levels | at 4 hours post-injection
  defined as the difference between the measurement at H8 and the measurement at H0 (4 hours prior to injection) of estradiol
change in AMH levels | at 4 hours post-injection
  defined as the difference between the measurement at H8 and the measurement at H0 (4 hours prior to injection) of AMH.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Catteau-Jonard, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandre, Lille, France